CLINICAL TRIAL: NCT00645723
Title: Phase 3b Randomized Double Blind Controled Placebo Comparative Trial of Intravenous Colistin vs Intravenous Colistin Plus Nebulized Colistin in Patients With Ventilator-associated Pneumonia (VAP) Due Multiresistant Acinetobacter Baumanii
Brief Title: Intravenous Colistin Versus Intravenous Colistin Plus Nebulized Colistin in VAP Due MDR Acinetobacter Baumannii
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: JOSÉ GARNACHO MONTERO, Servicio de Cuidados Críticos y Urgencias. Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COL\VAP
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Cross Infection; Pneumonia, Bacterial
Keywords: Acinetobacter baumanii; Ventilator-associated pneumonia
MeSH Terms: conditions — Cross Infection; Pneumonia, Bacterial; Pneumonia, Ventilator-Associated | interventions — Colistin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Intravenous colistin and nebulized colistin
  Interventions: Drug: Colistin
- B (Placebo Comparator): intravenous colistin and saline solution nebulized
  Interventions: Drug: Colistin and saline solution

INTERVENTIONS:
Drug: Colistin — intravenous colistin and nebulized colistin
  Arms: A
Drug: Colistin and saline solution — intravenous colistin and nebulized saline solution
  Arms: B

SUMMARY:
Compare the clinical efficiency evaluated by the treatment of the intravenous colistin plus inhaled colistin opposite to the treatment with colistin intravenous plus inhaled saline solution in patients with VAP due to baumannii carbapenems resistant.

DETAILED DESCRIPTION:
Compare the clinical efficiency evaluated by the treatment of the intravenous colistin plus inhaled colistin opposite to the treatment with colistin intravenous plus inhaled saline solution in patients with VAP due to baumannii carbapenems resistant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of VAP due A. baumannii or A. baumannii and another microorganism carbapenems resistant.
* Clinical Pulmonary Infection Score (CPIS) > 6

Exclusion Criteria:

* Allergy to colistin.
* Asthma
* Shock status
* Diagnose of VAP due A. baumannii colistin resistant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Compare the clinical efficiency evaluated by the treatment of the intravenous colistin plus inhaled colistin opposite to the treatment with colistin intravenous plus inhaled saline solution in patients with VAP due to baumannii carbapenems resistant | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Seville, Spain